CLINICAL TRIAL: NCT01837030
Title: Capsule Endoscopy Versus Conservative Therapy for Obscure Gastrointestinal Bleeding
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not feasible due to funding
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro00023612
Record Dates: First submitted 2013-04-04; First posted 2013-04-22 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Hemorrhage; Anemia
MeSH Terms: conditions — Hemorrhage; Anemia | interventions — ferrous sulfate; Capsule Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Oral Iron (Other)
  Interventions: Dietary Supplement: Ferrous sulfate
- Oral Iron and Capsule Endoscopy (Other)
  Interventions: Dietary Supplement: Ferrous sulfate; Device: Capsule Endoscopy

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate — Ferrous sulfate 325mg by mouth twice daily for the duration of the 12 month follow up period
Device: Capsule Endoscopy — GIVEN capsule
  Arms: Oral Iron and Capsule Endoscopy

SUMMARY:
This study is a single center prospective randomized control trial comparing the utility of performing capsule endoscopy compared to conservative management with oral iron therapy as the initial course of action in patients with non-severe obscure occult or obscure overt gastrointestinal (GI) bleeding. The investigators hypothesize that outcomes in patients with non-severe obscure GI bleeding who receive conservative therapy with oral iron will not differ to those on oral iron who undergo capsule endoscopy.

DETAILED DESCRIPTION:
Although the American Gastroenterological Association suggests that patients with obscure GI bleeding undergo a capsule endoscopy after a negative esophagogastroduodenoscopy (EGD) and colonoscopy, current recommendations from the British Society of Gastroenterology argue that unless there is an inadequate response to iron therapy, further imaging of the small bowel is probably not necessary. Several studies have demonstrated that this approach is reasonably safe. Furthermore, Laine et al demonstrated that when patients with obscure GI bleeding were randomized to either capsule endoscopy or dedicated small bowel contrast radiography, the rates of further bleeding, measured by subsequent hospitalization and blood transfusion events, were similar between the two groups. No study has randomized patients with obscure GI bleeding to receive capsule endoscopy vs. conservative therapy with oral iron.

This study is a single center prospective randomized control trial comparing the utility of performing capsule endoscopy compared to conservative management with oral iron therapy as the initial course of action in patients with non-severe obscure occult or obscure overt gastrointestinal bleeding. All patients will be recruited in the G.I. clinic, the endoscopy unit, or during inpatient consults after negative upper endoscopy and colonoscopy. The study will be explained to patients who qualify at that time. During this visit, patients will be questioned with regard to lower or upper G.I. symptoms, including abdominal pain, dyspepsia, nausea, vomiting, weight loss, diarrhea, change in stool character, melena and intermittent hematochezia. All patients will be started on standard dose oral iron therapy after informed consent. If the patient is already taking iron supplements, their dose with be adjusted to the standard regimen after informed consent. Patients will then be randomized to undergo capsule endoscopy or not. For patients randomized to undergo capsule endoscopy, all subsequent evaluation and treatment will be determined by capsule findings (i.e. capsule directed management) and standard of care at our institution.

Patients will be followed for 1 year. Follow up lab draws will occur at 1, 3, 6 and 12 months. They will consist of a complete blood count (CBC) and ferritin and can be performed at either the Medical University of South Carolina (MUSC) or an outside facility or office. If performed outside of MUSC, a standard medical records release form will be utilized to obtain the lab information. Patients will be provided with a paper card indicating their date of enrollment in the study. This card will be kept by the patient for the entire 12 month follow up period and will be collected at the end of the follow up period. The card will have an area where the patient can write the date of their first blood transfusion after enrollment. There will also be numerical checkboxes that the patient will check off for each unit of packed red blood cells (RBCs) they receive during the 12 month follow up period. Telephone calls will be made to each patient every 3 months after enrollment to inquire about hospitalizations and bleeding related procedures (including endoscopy, capsule, small bowel radiology, interventional radiology and surgery). Records of these hospitalizations and procedures will be obtained using a standard medical records release form.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and post-menopausal women with iron deficiency anemia and pre-menopausal women with iron deficiency anemia and a negative gynecologic workup or adults with overt GI bleeding as defined by melena or hematochezia with a ≥2 gram drop in hemoglobin after stabilization (Iron deficiency is defined as hemoglobin <13.7 g/dL in men and <12 g/dL in women with serum ferritin level <50 ng/mL). Also, patients with an otherwise unexplained drop in hemoglobin of ≥ 2 g/dL in the setting of hemoccult positive stool
* Negative EGD and colonoscopy for source of GI bleeding within six months of enrollment into the study.

Exclusion Criteria:

* Ongoing overt gastrointestinal bleeding requiring ≥4 units of packed RBC's on any given day in the setting of overt bleeding, blood transfusions on separate days (separated by ≥12 hours), or ≥6 units of packed RBC's over the previous 7-day period prior to presentation, in the setting of overt bleeding.
* Myocardial infarct, acute neurologic event, sepsis, or respiratory failure within the previous 1 week
* History of small bowel obstruction
* Pregnant women
* Prisoners
* Age less than 18
* Known GI or hematologic malignancy
* Achalasia
* Contraindications to capsule endoscopy (inability to take prep), or felt unsafe to undergo capsule as per study investigators
* Esophageal stricture that precludes even endoscopic capsule placement
* History of upper GI or small bowel surgery
* Inability to take oral iron.
* Active IV iron use.
* Alternate source of blood loss (e.g., menorrhagia)
* Hematemesis sufficient to be the cause of the hemoglobin decline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Time to first blood transfusion after randomization | 12 month follow up period
  Time-to-event analysis. Patients will be provided an index card on which they will record the date of their first blood transfusion after randomization

SECONDARY OUTCOMES:
Total number of blood transfusions | 3, 6, 9, and 12 months
Total number of hospitalizations | 3, 6, 9, and 12 months
Persistent Iron Deficiency Anemia as measured by ferritin and hemoglobin | 1, 3, 6, and 12 months
Total number of bleeding-related procedures performed after randomization | 3, 6, 9, and 12 months
Mortality | 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brock, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Goddard AF, James MW, McIntyre AS, Scott BB; British Society of Gastroenterology. Guidelines for the management of iron deficiency anaemia. Gut. 2011 Oct;60(10):1309-16. doi: 10.1136/gut.2010.228874. Epub 2011 May 11. PMID 21561874
- [Background] Gordon S, Bensen S, Smith R. Long-term follow-up of older patients with iron deficiency anemia after a negative GI evaluation. Am J Gastroenterol. 1996 May;91(5):885-9. PMID 8633576
- [Background] McLoughlin MT, Tham TC. Long-term follow-up of patients with iron deficiency anaemia after a negative gastrointestinal evaluation. Eur J Gastroenterol Hepatol. 2009 Aug;21(8):872-6. doi: 10.1097/MEG.0b013e328321836c. PMID 19282769
- [Background] Laine L, Sahota A, Shah A. Does capsule endoscopy improve outcomes in obscure gastrointestinal bleeding? Randomized trial versus dedicated small bowel radiography. Gastroenterology. 2010 May;138(5):1673-1680.e1; quiz e11-2. doi: 10.1053/j.gastro.2010.01.047. Epub 2010 Feb 2. PMID 20138043